CLINICAL TRIAL: NCT05738616
Title: Lenvatinib Combined With Transcatheter Arterial Chemoembolization and Camrelizumab Versus Lenvatinib Combined With Transcatheter Arterial Chemoembolization in Conversion Resection for Advanced Hepatocellular Carcinoma:A Randomized, Open-label, Parallel-controlled, Phase III Study(LEN-TAC Study)
Brief Title: Lenvatinib Combined With TACE and Camrelizumab in Conversion Resection for Advanced Hepatocellular Carcinoma (LEN-TAC Study)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Wen Tianfu (Other)
Responsible Party: Sponsor-Investigator, Wen Tianfu, Professor, West China Hospital
Organization: West China Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HX-IRB-AF-03-V1.0
Record Dates: First submitted 2023-02-12; First posted 2023-02-22 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: Conversion resection; Lenvatinib; Transcatheter arterial chemoembolization; Camrelizumab; Advanced hepatocellular carcinoma
MeSH Terms: interventions — camrelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lenvatinib combined with TACE and camrelizumab (Experimental)
  Interventions: Combination Product: Lenvatinib combined with TACE and Camrelizumab
- lenvatinib combined with TACE (Active Comparator)
  Interventions: Combination Product: Lenvatinib combined with TACE and Camrelizumab

INTERVENTIONS:
Combination Product: Lenvatinib combined with TACE and Camrelizumab — Once subjects have signed the informed consent and passed screening, they will be randomized in a 1:1 ratio to either the experimental arm (lenvatinib combined with TACE and camrelizumab) or the control arm (lenvatinib combined with TACE).

SUMMARY:
Compared to systemic therapy alone, conversion therapy is promising to improve the prognosis of patients with advanced hepatocellular carcinoma (HCC). Triple therapy (lenvatinib combined with transcatheter arterial chemoembolization and camrelizumab) may have significant efficacy in conversion therapy for patients with advanced HCC, but its safety and efficacy remain unknown. To address this, we have designed a randomized, open-label, parallel-controlled trial to evaluate the safety and efficacy of lenvatinib combined with transcatheter arterial chemoembolization and camrelizumab versus lenvatinib combined with transcatheter arterial chemoembolization in conversion resection for advanced HCC. Totally 196 patients with BCLC C stage HCC will be rigorously screened and included, and the primary endpoints of the study are overall survival. This study aims to provide valuable insights into new treatment strategies for advanced HCC.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 18 and 75 years.
2. Patients with HCC who strictly meet the criteria outlined in the Guidelines for the Diagnosis and Treatment of Hepatocellular Carcinoma (2022Edition), or those diagnosed by histopathology or cytology.
3. No prior anticancer therapy for HCC(Excluding patients who have received two or fewer TACE treatments).
4. ECOG PS score of 0-1.
5. Child-Pugh class A to B.
6. BCLC stage C Patients: tumor localized in one half of the liver with portal vein tumor thrombus (Vp1-Vp4 patients without contralateral portal vein tumor thrombus).
7. At least one radiographically measurable lesion according to mRECIST.
8. For HBsAg-positive patients, HBV-DNA < 2000 IU/ml (10^4 copies/ml) when undergoing PD-1 monoclonal antibody treatment; HCV RNA negative when HCV antibody is positive.
9. Adequate organ function based on laboratory test results.
10. Adequate blood pressure control with up to 3 antihypertensive agents, defined as BP ≤ 150/90 mmHg at screening with no changes in antihypertensive therapy within 1 week prior to Cycle 1/Day 1.
11. Patients expected to survive more than 3 months.
12. Not planning to become pregnant.

Exclusion Criteria:

1. Known intrahepatic cholangiocarcinoma, sarcomatoid HCC, mixed hepatocellular carcinoma, and fibrolamellar cell carcinoma.
2. Extrahepatic metastasis of HCC.
3. Diffuse HCC or intrahepatic tumor burden ≥ 50% (including contralateral portal vein tumor thrombus, superior mesenteric vein tumor thrombus, and inferior vena cava tumor thrombus).
4. Contraindications to TACE or epirubicin.
5. Known hypersensitivity to lenvatinib ingredients.
6. Known hypersensitivity to the active ingredient or excipients of Camrelizumab.
7. Presence of other malignancies.
8. Pregnancy, lactation, or unwillingness to use effective contraceptive measures.
9. Class II or higher myocardial ischemia or infarction, poorly controlled arrhythmia, cardiac insufficiency class III-IV, or LVEF < 50%.
10. Abnormal coagulation function or bleeding tendency.
11. History of psychiatric disorders or substance abuse.
12. HIV infection.
13. Allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
14. Active infection.
15. Poor compliance such as floating population.
16. Prior treatment with anti-PD-1, anti-PD-L1, or anti-PD-L2 agents.
17. Active autoimmune disease requiring systemic therapy within 2 years prior to the first dose.
18. Systemic glucocorticoid or immunosuppressive therapy within 7 days prior to the first dose.
19. Clinically uncontrolled pleural/peritoneal effusion.
20. Active chronic hepatitis B or C.
21. Vaccination with live vaccines within 30 days prior to the first dose.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2024-05-10 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 3-year
  Time from randomization to death (any cause).

SECONDARY OUTCOMES:
Adverse events | 2 years
  The occurrence of any hematological or non-hematological toxicity event (≥ class Ⅲ), including but not limited to impaired liver function, impaired hematological system, hypertension, diarrhea, proteinuria, hand-foot syndrome, etc. Severity of adverse events will be graded according to CTCAE v5.0.
Objective response rate | 2 years
  The percentage of patients achieving complete response and partial response among all patients. Response to treatment will be evaluated according to mRECIST.
Disease control rate | 2 years
  The percentage of patients with complete response, partial response and stable disease among all patients.
Event-free survival | 2 years
  Time from randomization to disease progression, local recurrence, distant metastasis, or death, whichever occurs first, assessed by mRECIST
Overall survival at 2 years | 2 years
  The time from start of treatment until death from any cause or the end of the study (the last enrolled patient should be followed for at least 2 years
Conversional resection rate | 2 years
  conversional resection patients/enrolled patients

CONTACTS AND LOCATIONS:
Locations (1):
- HuaXi hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided